CLINICAL TRIAL: NCT02487368
Title: Effects of a Mechanical Needle Stimulation Pad on Chronic Low Back Pain
Acronym: NRM_2009
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Siemens-Betriebskrankenkasse (Industry)
Responsible Party: Principal Investigator, Gustav Dobos, Principle Investigator, Universität Duisburg-Essen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRM_2009
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Low Back Pain; Recurrent Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Needle stimulation pad (Experimental): a self-administered treatment with a mechanical needle stimulation pad, a mechanical device to be used for 30 minutes daily for 14 days.
  Interventions: Device: Needle stimulation pad

INTERVENTIONS:
Device: Needle stimulation pad
  Other Names: Shakti mat, Bed of nails

SUMMARY:
The needle stimulation pad is a self-care device, which has been promoted for pain control and well-being. The aim of the study was to test the efficacy of the pad for chronic/recurrent low back pain treatment.

Patients with non-specific chronic or recurrent low back pain were selected from a large health insurance company database and advised to use the pad daily for two weeks; outcomes were assessed at baseline, weeks 2 and 14. Primary outcome measure was pain intensity at week 2; secondary outcome measures included the Oswestry disability index (ODI), health-related quality of life (SF-36), the fear avoidance beliefs questionnaire (FABQ), analgesic medication consumption and safety.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* chronic or recurrent low back pain in the past 12 months
* average pain intensity 4 out of 10 points

Exclusion Criteria:

* malignant back pain
* congenital deformities of the spine
* dystonia or other movement disorders
* spinal surgery within 12 months prior
* pregnancy
* dermatological diseases in the areas treated
* tendency for hemorrhages
* severe mental illness
* recent treatment with anticoagulation, corticoid medication, acupuncture

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity | day 14
  Visual analogue scale

SECONDARY OUTCOMES:
Pain intensity | Week 14
  Visual analogue scale
Oswestry Low Back Pain Disability Index | Day 14
Oswestry Low Back Pain Disability Index | Week 14
Short Form 36 Health Survey Questionnaire (SF-36) | Day 14
Short Form 36 Health Survey Questionnaire (SF-36) | Week 14
Fear Avoidance Beliefs Questionnaire (FABQ) | Day 14
Fear Avoidance Beliefs Questionnaire (FABQ) | Week 14
Experiences with the intervention | Day 14
  Open question: "please indicate observed changes"
Medication use | Day 14
  Use of medication, daily log
Number of any adverse events | Day 14
Pain intensity measured immediately after the application, visual analogue scale | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, Professor, Principal Investigator — University of Duisburg-Essen